CLINICAL TRIAL: NCT00168389
Title: A Study of the Safety and Efficacy of a New Treatment for Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 206207-010
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone 700 μg (Experimental): 700 µg Dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Interventions: Drug: Dexamethasone
- Dexamethasone 350 μg (Experimental): 350 µg Dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Interventions: Drug: Dexamethasone
- Sham (Sham Comparator): Sham posterior segment drug delivery system - needle-less drug delivery system without study medication not less than every 6 months for up to 36 months.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Dexamethasone — 350 µg or 700 µg dexamethasone posterior segment drug delivery system - injection into the vitreous cavity not less than every 6 months for up to 36 months.
  Other Names: Posurdex®; Ozurdex®
  Arms: Dexamethasone 350 μg; Dexamethasone 700 μg
Other: Sham — Sham posterior segment drug delivery system - needle-less drug delivery system without study medication not less than every 6 months for up to 36 months.
  Arms: Sham

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone for the treatment of diabetic macular edema.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older with diabetic macular edema;
* Decrease in visual acuity in at least one eye as a result of macular edema (20/50 or worse);
* Visual acuity in other eye no worse than 20/200

Key Exclusion Criteria:

* Known anticipated need for ocular surgery within first 12 months of study;
* History of glaucoma or current high eye pressure requiring more than 1 medication;
* Uncontrolled systemic disease;
* Known steroid-responder;
* Use of systemic steroids
* Use of Warfarin/Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2005-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (10):
- Inglewood, California, United States
- Westmead, New South Wales, Australia
- Toronto, Ontario, Canada
- Prague, Czechia
- Hamburg, Germany
- Tel Aviv, Israel
- Rockwell Center, Makati, Philippines
- Coimbra, Portugal
- Cape Town, South Africa
- Barcelona, Spain

REFERENCES:
- [Derived] Kozak I, Do DV, Lai H, Ogidigben MJ, Lopez FJ. Time-in-Range Analysis of Responses after Intravitreal Dexamethasone Therapy in Eyes with Diabetic Macular Edema. Ophthalmol Sci. 2025 May 26;5(5):100833. doi: 10.1016/j.xops.2025.100833. eCollection 2025 Sep-Oct. PMID 40688490
- [Derived] Valentim CCS, Lai H, Ogidigben MJ, Singh RP, Talcott KE. Baseline factors affecting diabetic macular oedema resolution after intravitreal dexamethasone implant treatment: post hoc analysis of the MEAD study. BMC Ophthalmol. 2025 Jul 9;25(1):403. doi: 10.1186/s12886-025-04208-3. PMID 40634898
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Yoon YH, Boyer DS, Maturi RK, Bandello F, Belfort R Jr, Augustin AJ, Li XY, Bai Z, Hashad Y; Ozurdex MEAD Study Group. Natural history of diabetic macular edema and factors predicting outcomes in sham-treated patients (MEAD study). Graefes Arch Clin Exp Ophthalmol. 2019 Dec;257(12):2639-2653. doi: 10.1007/s00417-019-04464-2. Epub 2019 Oct 25. PMID 31654188
- [Derived] Danis RP, Sadda S, Li XY, Cui H, Hashad Y, Whitcup SM. Anatomical effects of dexamethasone intravitreal implant in diabetic macular oedema: a pooled analysis of 3-year phase III trials. Br J Ophthalmol. 2016 Jun;100(6):796-801. doi: 10.1136/bjophthalmol-2015-306823. Epub 2015 Nov 18. PMID 26581718
- [Derived] Augustin AJ, Kuppermann BD, Lanzetta P, Loewenstein A, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Dexamethasone intravitreal implant in previously treated patients with diabetic macular edema: subgroup analysis of the MEAD study. BMC Ophthalmol. 2015 Oct 30;15:150. doi: 10.1186/s12886-015-0148-2. PMID 26519345

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Started | 163 | 166 | 165
Completed | 107 | 118 | 70
Not Completed | 56 | 48 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham | Total
Number analyzed (Participants) | 163 | 166 | 165 | 494
Age, Customized [Number; unit: Participants]
  <45 years | 4 | 5 | 7 | 16
  45 to 65 years | 89 | 97 | 95 | 281
  >65 years | 70 | 64 | 63 | 197
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 66 | 63 | 190
  Male | 102 | 100 | 102 | 304

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Best Corrected Visual Acuity (BCVA) Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Percentage of Patients | 22.1 | 18.7 | 13.3

2. Secondary Outcome: Average Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The average BCVA is calculated across study visits for each patient. A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, 39 Months
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Letters
  Baseline | 56.2 (10.5) | 55.9 (9.64) | 56.8 (8.66)
  Average Change from Baseline Over 39 Months | 4.1 (8.26) | 4.3 (8.49) | 1.9 (7.74)

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Letters
  Baseline | 56.2 (10.5) | 55.9 (9.64) | 56.8 (8.66)
  Change from Baseline at Month 39/Final Visit | 4.1 (13.89) | 5.0 (11.97) | 0.8 (11.89)

4. Secondary Outcome: Percentage of Patients With a BCVA Improvement of ≥10 Letters From Baseline in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Percentage of Patients | 38.7 | 34.3 | 23.0

5. Secondary Outcome: Average Change From Baseline in Retinal Thickness as Measured by Optical Coherence Tomography (OCT)
Description: OCT is a laser-based, noninvasive, diagnostic system that provides high-resolution, three-dimensional images of the retina from which retinal thickness can be measured. The average OCT retinal thickness is calculated across study visits for each patient. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, 39 Months
Population: Intent to Treat: all randomized patients with data at the time point
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 162 | 165 | 165
Microns
  Baseline | 436.7 (145.88) | 457.4 (158.09) | 468.7 (129.61)
  Average Change from Baseline Over 39 Months | -101.1 (119.17) | -103.9 (137.88) | -37.8 (103.96)

6. Secondary Outcome: 10th Percentile for Time to BCVA Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Shorter durations of time to improvement are best. The 10th percentile represents the first 10% of patients to reach a BCVA improvement of ≥15 letters from baseline in the study eye.
Time Frame: Baseline, 39 Months
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Days
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Days | 50 [21 to NA] | 51 [30 to NA] | 150 [NA to NA]

7. Secondary Outcome: Percentage of Patients With BCVA Improvement of ≥15 Letters From Baseline in the Study Eye at 3-month Intervals
Description: as for outcome 1
Time Frame: Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 21, Month 24, Month 27, Month 30, Month 33, Month 36, Month 39/Final Visit
Population: Intent to Treat: all randomized patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Number analyzed (Participants) | 163 | 166 | 165
Percentage of Patients
  Month 3 | 14.1 | 13.9 | 6.1
  Month 6 | 14.1 | 10.2 | 7.9
  Month 9 | 19.0 | 18.1 | 8.5
  Month 12 | 13.5 | 15.1 | 9.1
  Month 15 | 15.3 | 16.3 | 7.3
  Month 18 | 17.2 | 9.6 | 10.9
  Month 21 | 16.6 | 15.1 | 9.1
  Month 24 | 14.1 | 15.1 | 10.9
  Month 27 | 20.2 | 19.3 | 12.7
  Month 30 | 16.6 | 19.9 | 11.5
  Month 33 | 22.1 | 17.5 | 11.5
  Month 36 | 20.9 | 19.9 | 12.7
  Month 39/Final Visit | 22.1 | 18.7 | 13.3

ADVERSE EVENTS:
Description: The Safety Population included all treated patients and was used for adverse event (AE) and Serious Adverse Event (SAE) reporting.
Arm/Group | Dexamethasone 700 μg | Dexamethasone 350 μg | Sham
Serious Adverse Events (participants affected / at risk) | 52/160 | 52/165 | 34/164
Other Adverse Events (participants affected / at risk) | 153/160 | 162/165 | 124/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dexamethasone 700 μg (N=160) | Dexamethasone 350 μg (N=165) | Sham (N=164)
Cardiac Failure Congestive (Cardiac disorders) | 2 | 3 | 1
Atrioventricular Block Complete (Cardiac disorders) | 2 | 1 | 2
Coronary Artery Occlusion (Cardiac disorders) | 2 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1 | 2
Angina Unstable (Cardiac disorders) | 1 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 5 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 2 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 2 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 2
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 2 | 3 | 1
Cataract (Eye disorders) | 2 | 2 | 1
Cataract Subcapsular (Eye disorders) | 1 | 2 | 0
Vitreous Adhesions (Eye disorders) | 1 | 1 | 1
Angle Closure Glaucoma (Eye disorders) | 1 | 0 | 0
Anterior Chamber Fibrin (Eye disorders) | 1 | 0 | 0
Corneal Erosion (Eye disorders) | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Lens Dislocation (Eye disorders) | 1 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0
Open Angle Glaucoma (Eye disorders) | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Diabetic Retinal Oedema (Eye disorders) | 0 | 0 | 1
Pupillary Block (Eye disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal Fistula (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 2
Multi-Organ Failure (General disorders) | 2 | 0 | 0
Drug Intolerance (General disorders) | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Diabetic Foot Infection (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Infectious Peritonitis (Infections and infestations) | 1 | 0 | 0
Lung Abscess (Infections and infestations) | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Diabetic Gangrene (Infections and infestations) | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 1 | 1
Abscess of Salivary Gland (Infections and infestations) | 0 | 1 | 0
H1N1 Influenza (Infections and infestations) | 0 | 1 | 0
Pharyngeal Abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1
Localised Infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Chest Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ilium Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Chemical Eye Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Open Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Glucose Fluctuation (Investigations) | 1 | 0 | 0
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/102 | 2/100 | 2/102
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 3 | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 2 | 2 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1
Carotid Artery Occlusion (Nervous system disorders) | 1 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Muscle Spasticity (Nervous system disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 2 | 0
Renal Failure (Renal and urinary disorders) | 1 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Bladder Prolapse (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Intermittent Claudication (Vascular disorders) | 0 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone 700 μg (N=160) | Dexamethasone 350 μg (N=165) | Sham (N=164)
Intraocular Pressure Increased (Investigations) | 66 | 62 | 8
Cataract (Eye disorders) | 63 | 60 | 15
Conjunctival Haemorrhage (Eye disorders) | 37 | 53 | 17
Macular Oedema (Eye disorders) | 21 | 15 | 16
Cataract Subcapsular (Eye disorders) | 20 | 21 | 8
Vitreous Haemorrhage (Eye disorders) | 18 | 35 | 10
Hypertension (Vascular disorders) | 17 | 19 | 12
Conjunctivitis (Eye disorders) | 15 | 8 | 7
Nasopharyngitis (Infections and infestations) | 13 | 8 | 16
Conjunctival Hyperaemia (Eye disorders) | 12 | 18 | 9
Cataract Nuclear (Eye disorders) | 12 | 10 | 4
Eye Pain (Eye disorders) | 11 | 12 | 6
Retinal Haemorrhage (Eye disorders) | 11 | 11 | 7
Diabetic Retinopathy (Eye disorders) | 10 | 5 | 4
Macular fibrosis (Eye disorders) | 9 | 14 | 6
Posterior Capsule Opacification (Eye disorders) | 9 | 12 | 3
Dry Eye (Eye disorders) | 8 | 10 | 4
Vitreous Floaters (Eye disorders) | 8 | 4 | 2
Vitreous Detachment (Eye disorders) | 7 | 10 | 4
Visual Acuity Reduced (Eye disorders) | 6 | 11 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 6 | 10
Retinal Exudates (Eye disorders) | 4 | 7 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.